CLINICAL TRIAL: NCT02889757
Title: the Safety and Effect in TB Patients With NAC
Brief Title: The Protective Effect for Liver Organ in Patients With Anti-TB Drugs Using of Acetylcysteine (NAC)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shih-Lung Cheng, Associate Professor, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: T-6621
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Protective Effect in TB-DIH; TB-DIH Means: Drug Induced Liver Function Abnormalities
Keywords: tuberculosis; acetylcysteine; hepatotoxicity
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NAC 1200 mg (Experimental): patients with add NAC (600) 1# bid use per day during the study period
  Interventions: Drug: Acteylcysteine
- NAC 2400 mg (Experimental): patients with add NAC (600) 2# bid use per day during the study period
  Interventions: Drug: Acteylcysteine
- NAC 0 mg (Placebo Comparator): patients with add NAC (600) 0# (placebo) use per day during the study period
  Interventions: Drug: Acteylcysteine

INTERVENTIONS:
Drug: Acteylcysteine — randomized into three arms

SUMMARY:
Animal studies have shown that INH-RIF-induced oxidative injury can be prevented by supporting the cellular antioxidant defense mechanism by N-acetylcysteine (NAC). However, there are few published data and large sample sizes regarding the protective effect of NAC against hepatotoxicty induced by anti-TB drugs in humans, to our knowledge.

Therefore, the investigators designed a clinical trial with the aim to see whether NAC could protect against anti-TB drug-induced hepatotoxicity (DIH)

DETAILED DESCRIPTION:
Isoniazid (INH), rifampicin (RIF), and pyrazinamide (PZA), the first-line drugs used for tuberculosis (TB) chemotherapy, are associated with hepatotoxicity. A high rate of hepatotoxicity has been reported in some developing countries compared with advanced countries with a similar dose schedule. Sharifzadeh et al. reported an incidence of 27.7% in Iran. The reasons for this higher rate of hepatotoxicity are not completely clear. Ethnic variations, advanced age, female sex, alcoholism, underlying liver disease, acetylator phenotype, hepatitis B and C virus, HIV infection, extensive pulmonary parenchymal disease, and hypoalbuminemia have been observed to be the risk factors for the development of drug-induced hepatotoxicity (DIH) because of anti-TB treatment.

The mechanism of DIH induced by anti-TB treatment is not yet fully understood. Sodhi et al. proposed oxidative stress as one of the likely mechanisms for INH-RIF-induced hepatic injury. It is well established that by augmenting a cellular antioxidative defense system, especially nonprotein thiols, that is, glutathione (GSH), cells can be protected against oxidative injuries produced by various drugs and chemicals.

The study will be performed with randomized trial for assessment and protective effects over liver function in patients receiving anti-TB agents and using NAC.

ELIGIBILITY:
Inclusion Criteria:

1. new diagnosed to have tuberculosis
2. age >20 years -

Exclusion Criteria:

1. acute hepatitis in a previous one year
2. TB drugs induced urticaria or Steven-Johnson syndrome
3. life less than one year due to advanced cancer status
4. non-tuberculosis mycobacteria，NTM patients
5. HIV patients
6. patients can not cooperate
7. Allergic reaction for NAC

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
the incidence of DIH | during the 6 months treatment
  the rate for

SECONDARY OUTCOMES:
the incidence for other side effects | 6 months
  side effects including GI upset, blurred vision, neuropathy, renal organ damage

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No